CLINICAL TRIAL: NCT07236853
Title: The Effect of Hand Sewing Practices on Suturing Skills in Midwifery Students.
Brief Title: The Effect of Hand Sewing Practices on Suturing Skills
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melek Şen Aytekin (Other)
Responsible Party: Sponsor-Investigator, Melek Şen Aytekin, Research Assistant, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GaziosmanpasaU-EBE-MŞA-02
Record Dates: First submitted 2025-09-30; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Midwifery Education; Suture; Skill Performance
Keywords: midwifery education; Suture; skill

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the study, one of the researchers will provide suture training to the Hand Sewing Group. The other three researchers will not know which student belongs to which group. After the first researcher completes the training, the other three researchers will assess the suture skills of both the Hand Sewing Group and the Standard Training Group using the Objective Structured Assessment of Technical Skill (OSATS). After the data collection process is complete, the data will be transferred to SPSS by the researcher. Once the data is transferred to SPSS, the Hand Sewing Group will be assigned a code of X, and the Standard Training Group will be assigned a code of Y. The statistical analyst will not know which code belongs to which group. After the analysis is complete, the codes will be assigned their own names, and the results will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Education Group (No Intervention): This group received the standard training provided as part of the Normal Birth and Postpartum Period course. This training used an 80-slide PowerPoint presentation. The training was delivered in two 50-minute sessions. Surgical suture kits and sponges were used to demonstrate suturing skills.
- Hand Sewing Group (Experimental): This group received the standard training provided as part of the Normal Birth and Postpartum Period course. An 80-slide PowerPoint presentation was used for this training. The training was delivered in two 50-minute sessions. Surgical suture kits and sponges were used to demonstrate suture skills. Following the standard training, this group received hand suture exercises. Students in this group received instruction in hand suture exercises. Hand suture exercises were practiced with the group for a total of four days, one day apart. Hand suture exercises were demonstrated using fabric, sponge, and paper. Straight stitching and basting techniques were demonstrated.
  Interventions: Other: Hand Sewing Group

INTERVENTIONS:
Other: Hand Sewing Group — Students in this group will be trained in hand-sewing exercises and then be asked to work on sewing skills for one hour three days a week. Hand-sewing exercises will be demonstrated using fabric, sponge, and paper. Straight stitch and basting techniques will be demonstrated.
  Arms: Hand Sewing Group

SUMMARY:
The overall aim of this study was to evaluate the effects of hand-held suture exercises on non-locking continuous suture skills used in episiotomy repair in midwifery students. The study, conducted with a randomized, single-blind, controlled design, aimed to generate evidence of psychomotor skill transfer using Objective Structured Assessment of Technical Skills based performance scores and secondary indicators (time, number of errors, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Volunteers participating in the study,
* Those taking the Normal Birth and Postpartum Term course for the first time,
* Those who have not received suture training before,
* Third-year midwifery students

Exclusion Criteria:

* Students who are absent on the day the course is taught.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Structured Assessment of Technical Skills | All students will be asked to apply a simple running suture to the sponge after the intervention is completed. Evaluators will evaluate students using this form throughout the application (approximately 30 minutes).
  It will be used to assess simple running suture skills. The form will include a checklist and a global rating scale. Each general performance criterion is scored from 1 to 5. Each step includes ratings such as "Cannot do," "Can do with little assistance," and "Can do easily." Each scale is scored from 1 to 5.
  This means the total score can range from 4 to 20. High scores on the scale indicate a good level of general technical skill.
Continue sutur skill evaluation form | The researchers will monitor and complete the student's application as they complete it. The application will take approximately 30 minutes to complete. Students will be monitored throughout the process using this form (approximately 30 minutes).
  This form was created by researchers. It contains 10 items. The items are on a 3-point Likert-type scale, ranging from "performed" to "incorrect" or "incomplete." Participants receive 2 points for performing the skill, 1 point for incomplete performance, and 0 points for not performing or performing it incorrectly. The total score ranges from 0 to 20. Higher scores indicate successful implementation.
Episiotomy Skills Self-Efficacy Scale | It will be used as a pre-test 5 minutes after the standard training. It will be used as a post-test 5 minutes after students practice the simple running suture.
  The Episiotomy Skills Self-Efficacy Scale (ESSES), developed by Hadımlı et al. (2023), was used to assess participants' self-efficacy perceptions regarding episiotomy application and repair. The scale consists of 17 items on a 5-point Likert-type scale (1 = Strongly disagree - 5 = Strongly agree). A two-factor structure (application and repair) was identified in the development study and was reported to explain 63.4% of the total variance. Turkish validity and reliability analyses were conducted within the scope of the same study, and the Cronbach's alpha coefficient was reported as 0.94.
Perceived Learning Scale | It will be used as a pre-test 5 minutes after the standard training. It will be used as a post-test 5 minutes after students practice the simple running suture.
  The Perceived Learning Scale, developed by Rovai et al. (2009), was used to measure students' cognitive, affective, and psychomotor perceptions of learning. The scale was adapted into Turkish by Albayrak, Güngören, and Horzum (2014). The Turkish form consists of nine items, and items 2 and 7 are reverse-scored. The scale is scored on a 5-point Likert-type scale (1 = Strongly disagree - 5 = Strongly agree), with higher scores indicating a stronger perception of learning.
Clinical Skills Self-Efficacy Scale | It will be used as a pre-test 5 minutes after the standard training. It will be used as a post-test 5 minutes after students practice the simple running suture.
  The Learning Self-Efficacy Scale for Clinical Skills (L-SES), developed by Bayazit, Gonullu, and Dogan (2022) and adapted to Turkish for validity and reliability, was used to assess self-efficacy perceptions related to clinical skills. The scale has a 14-item, single-factor structure and uses a 5-point Likert-type scoring system. The Turkish version's Cronbach's alpha was reported as 0.94.
State-Trait Anxiety Inventory | It will be used as a pre-test 5 minutes after the standard training. It will be used as a post-test 5 minutes after students practice the simple running suture.
  The State-Trait Anxiety Inventory (STAI), developed by Spielberger et al. (1983), was used to measure participants' state and trait anxiety levels, along with a form adapted for Turkish by Öner and Le Compte (1985). Two subscales, each consisting of 20 items (STAI-1 = State Anxiety, STAI-2 = Trait Anxiety), are scored on a 4-point Likert-type scale. The total score is calculated by correcting for reverse items.

OTHER OUTCOMES:
Personal Information Form | It is filled out as a pre-test 5 minutes after the standard training.
  The Personal Information Form was prepared by the researcher in line with the literature to determine the socio-demographic characteristics of the students (age, education level, employment status, health insurance, parents' education status, parents' occupation, etc.). It consists of 10 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa Üniversitesi, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No